CLINICAL TRIAL: NCT05913895
Title: The Effect of Hydrogen Water in Oral Mucositis, Oral Frailty, Pain and Quality of Life in Head and Neck Cancer Patients After Therapy
Brief Title: The Effect of Hydrogen Water in Oral Mucositis in Head and Neck Cancer Patients After Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20230082
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer; Oral Mucositis; Pain; Quality of Life
Keywords: head and neck cancer; hydrogen water; cancer related symptom
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Pain | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrogen water (Experimental): At the end of cancer treatment (chemotherapy, radiotherapy, or Chemoradiotherapy), a hydrogen water gargle (dissolved for 12 hours or longer) was administered by the investigator or a researcher every Monday through Friday. The changes in six scales described above were tracked in the experimental and control groups on days 1 (T1), 3 (T2), 7 (T3), and 14 (T4) after the end of treatment.
  Interventions: Other: hydrogen water
- boiled water (Placebo Comparator): At the end of cancer treatment (chemotherapy, radiotherapy, or Chemoradiotherapy),boiled water gargle was administered by the investigator or a researcher every Monday through Friday. The changes in six scales described above were tracked in the experimental and control groups on days 1 (T1), 3 (T2), 7 (T3), and 14 (T4) after the end of treatment.
  Interventions: Other: hydrogen water

INTERVENTIONS:
Other: hydrogen water — To investigate whether the intervention of hydrogen water adjuvant therapy can improve oral mucositis, oral frailty, pain and Quality of Life with head and neck cancer who have received radiation therapy or combined chemotherapy.
  Other Names: boiled water

SUMMARY:
Inpatients or outpatients diagnosed with head and neck cancer who met the inclusion and exclusion criteria were referred to the co-investigator(Dr. Chih-Jen Huang and Dr. Hui-Ching Wang), who then personally explained to each participant, the purpose and conduct of the study, so that they all understood their rights and interests before giving a written consent.

DETAILED DESCRIPTION:
The study design was a randomized controlled trial and a longitudinal study with structured questionnaires (17-question basic information questionnaire、 The World Health Organization scale, WHO、NCI-CTCAE V5.0、Brief Pain Inventory-Taiwan、oral frailty checklist、European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-head & neck). The participants were randomly assigned to the experimental group (gargling with hydrogen water) and the control group (gargling with boiled water) by block randomization through a questionnaire administered by the investigator. At the end of cancer treatment (chemotherapy, radiotherapy, or Chemoradiotherapy), a hydrogen water gargle (dissolved for 12 hours or longer) or boiled water gargle was administered by the investigator or a researcher every Monday through Friday. The changes in six scales described above were tracked in the experimental and control groups on days 1 (T1), 3 (T2), 7 (T3), and 14 (T4) after the end of treatment. The data from these scales were entered into a computer and analyzed using statistical software, and the overall data are presented to demonstrate the efficacy of hydrogen water.

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosed with head and neck cancer
2. adults over the age of 20
3. have normal cognition
4. can use Mandarin or Taiwanese to communicate
5. received radiation therapy or combined chemotherapy

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 2, 3 and 4
2. received oral cancer surgery within two months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-24 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0,Change From Baseline in Pain Scores on the Brief Pain Inventory-Taiwan Scale at 2 Weeks | 2 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Huang, Study Chair — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No